CLINICAL TRIAL: NCT00126009
Title: A 3-Month, Open, Randomised Trial Comparing the Efficacy and Safety of the Association Valproate-Amisulpride to the Association Valproate-Haloperidol in Bipolar I Patients Suffering From a Manic Episode
Brief Title: SOLMANIA - Comparison of Valproate-Amisulpride and Valproate-Haloperidol in Bipolar I Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C_8428
Record Dates: First submitted 2005-07-18; First posted 2005-08-02 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Amisulpride

INTERVENTIONS:
Drug: Amisulpride

SUMMARY:
The primary objective is:

* To compare the efficacy of the association valproate-amisulpride (400 to 800 mg/day) to the association valproate-haloperidol (5 to 15 mg/day) in bipolar I patients suffering from a manic episode according to DSM IV TR (American Psychiatric Association [APA] 2000) and treated for a 3-month period.

The secondary objectives are:

* To evaluate the clinical and biological safety of the association valproate-amisulpride to the association valproate-haloperidol;
* To assess the patient status 3 weeks and 3 months after inclusion; and
* To assess patient satisfaction at 3 months.

ELIGIBILITY:
Inclusion Criteria:

Pre-Inclusion Criteria on D-3:

* In-patients
* From 18 to 65 years old
* Able to comply with the protocol
* Having given their written informed consent (with a legal representative or a person of trust)
* Current diagnosis of bipolar I disorder according to DSM IV TR (APA 2000)
* Having had at least one manic episode in the past
* Currently suffering from a manic episode according to DSM IV TR (APA 2000)
* A minimum total score of 20 on the Young Mania Rating Scale (Y-MRS) at D-3

Inclusion Criteria on D0:

* Having completed at least one day of the one to three-day washout period
* A minimum total score of 20 on the Young Mania Rating Scale at D0
* A score of > or = 3 for 2 of the following Y-MRS items: elevated mood; increased motor activity energy; sleep; content (grandiosity).
* A score of > or = 5 on the Clinical Global Impression Severity Scale for the severity of mania items at D0
* Using an effective contraception method (women of childbearing age only)

Exclusion Criteria:

Exclusion Criteria on D-3:

* Having participated in a clinical trial within the three previous months
* Pregnant or breast-feeding. Female patients should therefore be using reliable contraceptive methods (oral or parenteral contraception, intra-uterine device or surgical sterilisation)
* Uncontrolled gastro-intestinal, renal, hepatic, endocrine, cardiovascular, pulmonary, immunological or hematological disease
* Central nervous system (CNS) neoplasm; demyelinating disease; degenerative neurological disorder; active CNS infection; or any progressive disorder that may confound interpretation of the study results
* Prolactin-dependant tumor
* Past or current pancreatitis
* Acute hepatitis, chronic hepatitis, or family history of severe hepatitis, especially drug related, hepatic porphyry
* Current or recent (within 3 months) DSM IV diagnosis of substance dependence (with the exception of nicotine or caffeine dependence); or substance abuse with stimulants including, but not limited to, cocaine, crack, amphetamines, pseudoephedrine, cold medications with phenylephrine, or other stimulants. Alcohol and marijuana abuse prior to study entry would be acceptable if related to the current manic episode, based on the investigator's judgement
* Parkinson's disease
* Phaeochromocytoma
* History of epilepsy
* History of allergy or hypersensitivity to haloperidol or benzamides or valproate
* Treated with fluoxetin within the past 4 weeks
* Treated with injectable long-acting neuroleptics if, for the patient, the interval between 2 injection periods has not elapsed before pre-inclusion (D-3)
* Treated with a mood stabiliser (other than valproate) at effective dose for less than 7 days preceding D-3 and for whom a modification is not justified
* Bradycardia < 55 beats per minute (bpm)
* Known hypokaliaemia
* Congenital prolongation of the QT interval
* Treated with any of the following medications: Class Ia antiarrhythmic agents such as quinidine, disopyramide/Class III antiarrhythmic agents such as amiodarone, sotalol; Drugs like: beperidil, cisapride, sultopride, thioridazine, intravenous (IV) erythromycin, IV vincamine, halofantrine, pentamidine, or sparfloxacin.

Exclusion Criteria on D0:

* Potentially significant alterations of laboratory tests on D0:

  * ASAT or ALAT > 2 upper limit of normal (ULN). If ASAT or ALAT values range between 1.5 ULN and 2 ULN, the patient can be randomized and a new test will be performed 7 days after randomization;
  * Alkaline phosphatase levels or bilirubin levels not within normal reference range.
* QTc prolongation on D0; QTc Bazett > 450ms in male patients and QTc > 470ms in female patients on electrocardiogram (ECG).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-05

PRIMARY OUTCOMES:
Combination of the percentage of responders defined by a decrease of at least 50% of the Y-MRS (Young Mania Rating Scale) between D0 and D END and the completion of the 3-month treatment period.

SECONDARY OUTCOMES:
Other efficacy criteria (such as the changes in Y-MRS scores between D0 and D 21, between D0 and D END.The percentage of remission defined as the Y-MRS < or = 12 at D END...). Safety data (clinical, ECG and laboratory data)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, MD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Bratislava, Slovakia
- Sanofi-Aventis, Barcelona, Spain